CLINICAL TRIAL: NCT07324954
Title: Impact of Irrigation Volumes in Revision Total Knee Arthroplasty (TKA) Surgical Washout: A Pilot Study
Brief Title: Methylene Blue in Total Knee Arthroplasty (TKA)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Colin A. McNamara, Assistant Professor of Orthopaedic Surgery, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20250901
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Total Knee Arthroplasty; Prosthetic-joint Infection; Irrigation
MeSH Terms: interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Revision Arthroplasty with Documented PJI (DAIR) (Experimental): Participants undergoing revision total knee arthroplasty for periprosthetic joint infection will receive standard of care revision surgery. During the procedure, methylene blue dye will be applied intra-articularly via soaked gauze to simulate contaminant presence. Irrigation will be performed in 2,000 mL increments until macroscopic clearance is achieved, documented intraoperatively.
  Interventions: Drug: Methylene Blue 10 MG/ML (intra-articular application); Procedure: Revision Arthroplasty for PJI (DAIR)
- Primary Total Knee Arthroplasty (Active Comparator): Participants undergoing primary total knee arthroplasty will receive standard of care primary surgery. During the procedure, methylene blue dye will be applied intra-articularly via soaked gauze to simulate contaminant presence. Irrigation will be performed in 2,000 mL increments until macroscopic clearance is achieved, which will be documented intraoperatively.
  Interventions: Drug: Methylene Blue 10 MG/ML (intra-articular application); Procedure: Primary Total Knee Arthroplasty

INTERVENTIONS:
Drug: Methylene Blue 10 MG/ML (intra-articular application) — 10 mL of 0.25% methylene blue dissolved in 20 mL normal saline, applied intra-articularly via sterile gauze to simulate contaminant presence. Irrigation performed in 2,000 mL increments until macroscopic dye clearance is achieved. Used solely as a surrogate marker; no therapeutic intent
Procedure: Revision Arthroplasty for PJI (DAIR) — Standard of care surgical procedure performed for documented periprosthetic joint infection
  Arms: Revision Arthroplasty with Documented PJI (DAIR)
Procedure: Primary Total Knee Arthroplasty — Standard of care surgical procedure performed for severe knee osteoarthritis
  Arms: Primary Total Knee Arthroplasty

SUMMARY:
The purpose of this pilot study is to determine the volume of irrigation required to achieve macroscopic clearance of contaminants during a debridement, antibiotics, and implant retention (DAIR) procedure for periprosthetic joint infection (PJI) of the knee. Given the lack of robust data guiding irrigation volume in this setting, the investigator proposes to use the application of methylene blue dye intraoperatively to simulate contaminant presence. Serial irrigation will be performed, with photographic documentation taken every 2,000mL until visible dye clearance is achieved. This study aims to identify the irrigation volumes that result in gross clearance of simulated contamination, thereby informing the design and stratification of a future randomized controlled trial (RCT) evaluating irrigation strategies in DAIR procedures.

ELIGIBILITY:
Inclusion Criteria:

* Primary Total Knee Arthroplasty (TKA) or Primary Total Knee Arthroplasty (TKA) with Prosthetic Joint Infection (PJI)
* 18 years
* Able to provide informed consent

Exclusion Criteria:

* Incomplete irrigation documentation
* Patients with severe immunosuppression (example: chemotherapy, neutropenia, Human Immunodeficiency Virus [HIV], steroid use)
* Positive fungal, parasitic, or mycobacterial cultures
* Methylene Blue allergy
* Patients on Monoamine Oxidase (MAO) inhibitors, Selective Serotonin Reuptake Inhibitors (SSRI), Selective Norepinephrine Reuptake Inhibitors (SNRI), and/or Tricyclic Antidepressants (TCA)
* History of methemoglobinemia
* Glucose-6-Phosphate (G6P) Enzyme Deficiency
* Chronic Kidney disease or Glomerular Filtration Rate (GFR) less than 30mL/min
* Prisoners
* Pregnant Woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Irrigation Volume Required for Clearance of Methylene Blue Dye | Within 15 minutes intraoperatively, immediately following methylene blue dye application and completion of irrigation procedure
  To determine the volume of irrigation fluid (mL) required to achieve complete macroscopic clearance of methylene blue dye from the surgical site. The irrigation volume will be recorded intraoperatively at each increment and clearance assessed by direct visual confirmation

CONTACTS AND LOCATIONS:
Overall Officials: Colin A McNamara, MD, MBA, Principal Investigator — University of Miami
Locations (1):
- UHealth Tower, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No